CLINICAL TRIAL: NCT04329962
Title: Comparison of Bioavailability and Urinary Metabolite Profile After Consumption of Blueberry Extract and Whole Blueberry Powder Confections in Healthy Men and Women
Brief Title: Metabolism and Absorption of Anthocyanins From Extract and Whole Blueberry Powder Confections in Healthy Adults
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Principal Investigator, Yael Vodovotz, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: OSU-18010; NCI-2020-01525 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2020-03-25; First posted 2020-04-01 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Healthy Diet; Nutrition Aspect of Cancer
MeSH Terms: interventions — Diet Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group I (blueberry extract, blueberry powder) (Experimental): Participants undergo a washout on days -7 to -1 and then consume blueberry extract confection on day 0. Participants undergo a second washout on days 1-7 and then consume blueberry powder confection on day 8.
  Interventions: Other: Blueberry Powder Food Product; Other: Dietary Intervention; Other: Questionnaire Administration
- Group II (blueberry powder, blueberry extract) (Experimental): Participants undergo a washout on days -7 to -1 and then consume blueberry powder confection on day 0. Participants undergo a second washout on days 1-7 and then consume blueberry extract confection on day 8.
  Interventions: Other: Blueberry Powder Food Product; Other: Dietary Intervention; Other: Questionnaire Administration

INTERVENTIONS:
Other: Blueberry Powder Food Product — Consume blueberry powder confection
Other: Dietary Intervention — Consume blueberry extract confection
  Other Names: Dietary Modification; intervention, dietary; Nutrition Intervention; Nutrition Interventions; Nutritional Interventions
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This trial studies how well a group of compounds found in blueberries called anthocyanins are absorbed into the body from 2 different types of blueberry confections (blueberry extract and whole blueberry powder). Blueberries contain several compounds which may be beneficial for human health and prevention of disease. These compounds can be consumed as part of a complex matrix in the whole fruit or also in a simplified matrix in the form of a fruit extract. Studying the absorption and metabolism of these compounds may help researchers understand how they influence health and disease, as well as determining the role of the food matrix on absorption of berry phytochemical.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Compare urinary flavonoids composition, compliance and sensory acceptability of 2 blueberry-based amorphous functional confections one containing blueberry extract and the other of a whole blueberry powder) formulated to deliver the 320 mg of anthocyanins.

II. Assess the effect of blueberry source (extract versus [vs] whole fruit powder) on urinary metabolomics profile.

OUTLINE: Participants are randomized to of 2 groups.

GROUP I: Participants undergo a washout on days -7 to -1 and then consume blueberry extract confection on day 0. Participants undergo a second washout on days 1-7 and then consume blueberry powder confection on day 8.

GROUP II. Participants undergo a washout on days -7 to -1 and then consume blueberry powder confection on day 0. Participants undergo a second washout on days 1-7 and then consume blueberry extract confection on day 8.

ELIGIBILITY:
Inclusion Criteria:

* Be healthy, free-living adults
* Have a body mass index (BMI) between 18 and 35 kg/m^2
* Be a non-smoker (defined as adults who have never smoked or who have not had a cigarette in the past ten years)
* Agree to follow a berry-restricted diet and to document any accidental consumption of restricted foods each day of the study

Exclusion Criteria:

* Report being actively treated for any metabolic, digestive or immunologic disorder including malabsorptive disorders, renal insufficiency, hepatic insufficiency, any autoimmune disorder or short bowel syndrome
* Have a known allergy or food intolerance to ingredients in study products (blueberries), other berries, wheat, or soy
* Are strict vegans (no consumption of animal, fish or egg products)
* Are planning to conceive, or are currently pregnant or lactating
* Are heavy alcohol consumers (defined as an average consumption of greater than 2 drinks/ day)
* Have been on an antibiotic regime lasting for one week in the last 6 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2018-05-08 (Actual); Primary Completion 2018-05-14 (Actual); Study Completion 2026-07-10 (Estimated)

PRIMARY OUTCOMES:
Acceptability | Day 0 of each arm
  Means +/- SD (standard deviation) will be used to express the results from acceptability tests, and differences in acceptability of the two confections will be determined using paired t tests using the SPSS statistical software package.
Acceptability | Day 8 of each arm
  Means +/- SD (standard deviation) will be used to express the results from acceptability tests, and differences in acceptability of the two confections will be determined using paired t tests using the SPSS statistical software package.
Bioavailability of the various berry interventions | Day 1 of each arm
  Will measure bioavailability of the various berry interventions using high performance liquid chromatography (HPLC) analysis of blueberry phytochemicals and metabolites in urine at the day 1 timepoint, after consumption of the test product. Baseline comparisons for anthocyanins found in urine between trials will be performed a paired t-test. Total anthocyanins in 24-hour urine after consumption of one blueberry treatment will be compared to each participant's baseline urine and to total anthocyanins after consumption of the blueberry treatment in a paired t-test.
Bioavailability of the various berry interventions | Day 8 of each arm
  Will measure bioavailability of the various berry interventions using high performance liquid chromatography (HPLC) analysis of blueberry phytochemicals and metabolites in urine at the day 8 timepoints. Baseline comparisons for anthocyanins found in urine between trials will be performed a paired t-test. Total anthocyanins in 24-hour urine after consumption of one blueberry treatment will be compared to each participant's baseline urine and to total anthocyanins after consumption of the blueberry treatment in a paired t-test.

CONTACTS AND LOCATIONS:
Overall Officials: Yael Vodovotz, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu